CLINICAL TRIAL: NCT04682483
Title: Cardiogenic Shock Working Group Registry
Acronym: CSWG
Status: Recruiting | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Abbott (Industry); Boston Scientific Corporation (Industry); Abiomed Inc. (Industry); Getinge Group (Other)
Responsible Party: Sponsor
Other Study IDs: 12670
Record Dates: First submitted 2020-12-07; First posted 2020-12-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic Shock; mechanical circulatory support; hemodynamics; heart failure; acute myocardial infarction; registry; critical care; clinical outcomes research
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardiogenic Shock Patients: Cardiogenic Shock patients eligible for this study are defined by at least one of the two categories below.
  1. Patients have at least 2 of the following concurrently at any point during the index hospitalization: MAP < 60mmHg or a >30mmHg drop in MAP from baseline, SBP < 90mmHg or a >30mmHg drop in SBP from baseline, Pulse > 100, Cardiac Index < 2.2, Cardiac Power Output ≤ 0.6 or PAPI < 1.0.
  2. Patients require the use of at least 1 vasopressor, inotrope or acute mechanical circulatory support device to maintain values above the above targets.
  Interventions: Drug: Vasopressor; Drug: Inotrope; Device: Acute Mechanical Circulatory Support Devices

INTERVENTIONS:
Drug: Vasopressor — The vasopressors include phenylephrine, norepinephrine, epinephrine, dopamine and vasopressin.
Drug: Inotrope — Inotropes include dobutamine and milrinone.
Device: Acute Mechanical Circulatory Support Devices — Acute Mechanical Circulatory Support devices include ECMO (VV), ECMO (VA), Impella CP, Impella 2.5, Impella 5.0, Impella 5.5, Impella RP, IABP, Centrimag, Tandem Heart and ProTek Duo.

SUMMARY:
The Cardiogenic Shock Working Group is a multicenter registry where we collect de-identified clinical variables from the medical records and follow-up phone calls of shock patients from multiple institutions and centralize this data to a single registry for analysis of clinical outcomes.

DETAILED DESCRIPTION:
The Cardiogenic Shock Working Group is an Academic Research Consortium involving multiple medical centers within the United States and includes a multicenter registry for patients with cardiogenic shock. De-identified clinical variables are collected from medical records and follow-up phone calls. There is currently no central database for cardiogenic shock, therefore analysis of cardiogenic shock on a larger scale is limited. A goal of the Cardiogenic Shock Working Group is to create a centralized registry, compiled of data from multiple institutions, to analyze clinical outcomes. The Cardiogenic Shock Working Group Registry will include a retrospective arm, where data is collected during the course of the hospital stay, and a prospective arm, where long-term outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cardiogenic shock.

Cardiogenic shock is defined by at least one of the two categories below:

1. At least 2 of the following concurrently at any point during the index hospitalization:

   * Cardiac Index < 2.2
   * PAPI < 1.0
   * Cardiac Power Output ≤ 0.6
   * MAP < 60mmHg or a >30mmHg drop in MAP from baseline
   * SBP < 90mmHg or a >30mmHg drop in SBP from baseline
   * Pulse > 100
2. Require at least one acute mechanical circulatory support device, vasopressor or inotrope to maintain values above the above target.

Post-cardiotomy patients must meet the inclusion criteria 72 hours after their surgery to be included in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are 18 or older who have an official diagnosis of cardiogenic shock.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Mortality | 30 days after discharge
  Death in subjects during the time frame.
Rate of Mortality | 1 year after discharge
  Death in subjects during the time frame.

SECONDARY OUTCOMES:
Rate of Re-hospitalization | 30 day after discharge
  We will be observing if patient was hospitalized again during the 1 year-time frame. We will collect information on surgeries and interventions during the course of rehospitalization.
Rate of Re-hospitalization | 1 year after discharge
  We will be observing if patient was hospitalized again during the 1 year-time frame. We will collect information on surgeries and interventions during the course of rehospitalization.
New York Heart Association (NYHA) Class | 30 day after discharge
  NYHA Classification provides a way to classify the stages of heart failure. Class I- No symptoms and no limitation in ordinary physical activity Class II- Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity Class IV - Severe limitations
New York Heart Association (NYHA) Class | 1 year after discharge
  NYHA Classification provides a way to classify the stages of heart failure. Class I- No symptoms and no limitation in ordinary physical activity Class II- Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity Class IV - Severe limitations

CONTACTS AND LOCATIONS:
Overall Officials: Reshad Garan, MD, Study Director — Beth Israel Deaconess Medical Center; Claudius Mahr, DO, Study Director — University of Washington; Jaime Hernandez-Montfort, MD, Study Director — Cleveland Clinic Foundation-Florida; Daniel Burkhoff, MD PhD, Study Director — CardioVascular Research Foundation
Locations (16):
- United States (16):
  - Cleveland Clinic Florida, Weston, Florida
  - Northwestern Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Providence St. Vincent Heart Clinic, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Scott & White Advanced Heart Failure Clinic, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Inova Health System, Falls Church, Virginia
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapur NK, Thayer KL, Zweck E. Cardiogenic Shock in the Setting of Acute Myocardial Infarction. Methodist Debakey Cardiovasc J. 2020 Jan-Mar;16(1):16-21. doi: 10.14797/mdcj-16-1-16. PMID 32280413
- [Background] Pahuja M, Chehab O, Ranka S, Mishra T, Ando T, Yassin AS, Thayer KL, Shah P, Kimmelstiel CD, Salehi P, Kapur NK. Incidence and clinical outcomes of stroke in ST-elevation myocardial infarction and cardiogenic shock. Catheter Cardiovasc Interv. 2021 Feb 1;97(2):217-225. doi: 10.1002/ccd.28919. Epub 2020 Apr 30. PMID 32352638
- [Background] Thayer KL, Zweck E, Ayouty M, Garan AR, Hernandez-Montfort J, Mahr C, Morine KJ, Newman S, Jorde L, Haywood JL, Harwani NM, Esposito ML, Davila CD, Wencker D, Sinha SS, Vorovich E, Abraham J, O'Neill W, Udelson J, Burkhoff D, Kapur NK. Invasive Hemodynamic Assessment and Classification of In-Hospital Mortality Risk Among Patients With Cardiogenic Shock. Circ Heart Fail. 2020 Sep;13(9):e007099. doi: 10.1161/CIRCHEARTFAILURE.120.007099. Epub 2020 Sep 9. PMID 32900234
- [Background] Whitehead E, Thayer K, Kapur NK. Clinical trials of acute mechanical circulatory support in cardiogenic shock and high-risk percutaneous coronary intervention. Curr Opin Cardiol. 2020 Jul;35(4):332-340. doi: 10.1097/HCO.0000000000000751. PMID 32487943
- [Background] Kapur NK, Whitehead EH, Thayer KL, Pahuja M. The science of safety: complications associated with the use of mechanical circulatory support in cardiogenic shock and best practices to maximize safety. F1000Res. 2020 Jul 29;9:F1000 Faculty Rev-794. doi: 10.12688/f1000research.25518.1. eCollection 2020. PMID 32765837
- [Background] Garan AR, Kanwar M, Thayer KL, Whitehead E, Zweck E, Hernandez-Montfort J, Mahr C, Haywood JL, Harwani NM, Wencker D, Sinha SS, Vorovich E, Abraham J, O'Neill W, Burkhoff D, Kapur NK. Complete Hemodynamic Profiling With Pulmonary Artery Catheters in Cardiogenic Shock Is Associated With Lower In-Hospital Mortality. JACC Heart Fail. 2020 Nov;8(11):903-913. doi: 10.1016/j.jchf.2020.08.012. PMID 33121702
- [Background] Whitehead EH, Thayer KL, Burkhoff D, Uriel N, Ohman EM, O'Neill W, Kapur NK. Central Venous Pressure and Clinical Outcomes During Left-Sided Mechanical Support for Acute Myocardial Infarction and Cardiogenic Shock. Front Cardiovasc Med. 2020 Aug 28;7:155. doi: 10.3389/fcvm.2020.00155. eCollection 2020. PMID 33005634
- [Background] Pahuja M, Ranka S, Chehab O, Mishra T, Akintoye E, Adegbala O, Yassin AS, Ando T, Thayer KL, Shah P, Kimmelstiel CD, Salehi P, Kapur NK. Incidence and clinical outcomes of bleeding complications and acute limb ischemia in STEMI and cardiogenic shock. Catheter Cardiovasc Interv. 2021 May 1;97(6):1129-1138. doi: 10.1002/ccd.29003. Epub 2020 May 30. PMID 32473083
- [Derived] Hernandez-Montfort J, Kanwar M, Sinha SS, Garan AR, Blumer V, Kataria R, Whitehead EH, Yin M, Li B, Zhang Y, Thayer KL, Baca P, Dieng F, Harwani NM, Guglin M, Abraham J, Hickey G, Nathan S, Wencker D, Hall S, Schwartzman A, Khalife W, Li S, Mahr C, Kim J, Vorovich E, Pahuja M, Burkhoff D, Kapur NK. Clinical Presentation and In-Hospital Trajectory of Heart Failure and Cardiogenic Shock. JACC Heart Fail. 2023 Feb;11(2):176-187. doi: 10.1016/j.jchf.2022.10.002. Epub 2022 Oct 31. PMID 36342421
- [Derived] Kapur NK, Kanwar M, Sinha SS, Thayer KL, Garan AR, Hernandez-Montfort J, Zhang Y, Li B, Baca P, Dieng F, Harwani NM, Abraham J, Hickey G, Nathan S, Wencker D, Hall S, Schwartzman A, Khalife W, Li S, Mahr C, Kim JH, Vorovich E, Whitehead EH, Blumer V, Burkhoff D. Criteria for Defining Stages of Cardiogenic Shock Severity. J Am Coll Cardiol. 2022 Jul 19;80(3):185-198. doi: 10.1016/j.jacc.2022.04.049. PMID 35835491